CLINICAL TRIAL: NCT06711536
Title: Evaluating the Trauma and Injury Severity Score (TRISS) as a Predictor of Patient Outcomes: A Prospective Observational Study in the Trauma and Emergency Department of Al-Kadhimiya Teaching Hospital, Iraq
Brief Title: TRISS as a Predictor of Trauma Patient Outcomes
Acronym: TRISS/ER
Status: Recruiting | Type: Observational
Sponsor: Al-Nahrain University (Other)
Responsible Party: Principal Investigator, Abdul-Ilah R. Khamis, Principal Investigator, Al-Nahrain University
Other Study IDs: UNCOMIRB20241134
Record Dates: First submitted 2024-11-23; First posted 2024-12-02 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Trauma, Multiple
Keywords: TRISS
MeSH Terms: conditions — Multiple Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of this prospective observational study is to evaluate the predictive utility of the Trauma and Injury Severity Score (TRISS) in determining patient outcomes, including survival and mortality, among trauma patients admitted to the trauma and emergency department of Kadhimiya Educational Hospital, Iraq.

The main questions it aims to answer are:

How accurately does TRISS predict survival and mortality outcomes in trauma patients? What is the performance of TRISS in predicting secondary outcomes, such as the need for intensive care, surgical interventions, and length of hospital stay?

Participants will:

Be assessed using the TRISS score upon their admission to the emergency department.

Have their clinical outcomes, including survival, need for intensive care, surgery, and hospital stay, monitored throughout their hospitalization.

DETAILED DESCRIPTION:
Trauma is a significant cause of mortality and morbidity around the world. Approximately 10% of the burden of disease in adults is due to traumatic injuries. Trauma can lead to serious consequences, including disabilities, psychosocial burdens, and increased mortality among the actively working population. Cardiopulmonary arrest, unplanned admissions to intensive care units, and nosocomial infections are some complications faced by trauma patients admitted to trauma centers. The estimated mortality rate for hospitalized trauma patients is 11%. The in-hospital mortality rate for trauma patients who undergo cardiopulmonary resuscitation (CPR) is 92.7%. Trauma-related mortality and morbidity depend on injury severity, diagnostic delays, and the time taken to reach a medical facility.Timely evaluation, effective post-trauma care, and appropriate triage can significantly reduce long-term mortality and morbidity among trauma patients, with rapid assessment of trauma severity being crucial for the primary triage of multiple trauma patients.

Trauma scoring systems are valuable tools for quickly assessing the severity of injuries and predicting patient outcomes. By utilizing these scoring systems, healthcare providers can enhance the organization of trauma patient triage, optimize resource allocation, and conduct immediate evaluations of potential complications. Several scoring systems have been developed to assess trauma cases. These trauma scores are classified into three categories: anatomical (such as the Abbreviated Injury Scale and Injury Severity Score), physiological (like the Revised Trauma Score), and combined (such as the Trauma and Injury Severity Score). Physiological scores can be determined during the initial clinical assessment of the patient, while anatomical scoring can be performed later after the patient has been stabilized. This makes it easier to stratify trauma patients effectively. On the other hand, combined scores that include both anatomical and physiological criteria are more useful for patient prognosis. One such combined score is the Trauma and Injury Severity Score (TRISS), which was designed by the Major Trauma Outcome Study (MTOS) in the United States to predict the outcome in polytrauma patients and includes the Injury Severity Score (ISS) and Revised Trauma Score (RTS).

Trauma is thus now a significant health challenge in Iraq. Through the long fight in Iraq, more and more people are experiencing violence-related injuries, such as from firearms and attacks. The work also demonstrates that violence is one of the primary determinants of public health because it leads to complications with injuries and the psychological development of the survivors in the course of their lives. The Iraqi healthcare system has documented a significant rise in RTAs (road traffic accidents), particularly since the escalation of conflict around 2013. Trauma care system is not well established, and few protocols are followed clinically, and no scientific method is well established to predict the outcome in trauma patients in Iraq. This is made worse by scarce resources, inadequate staffing and educational preparedness of medical personnel, and the overall lack of formalized trauma registry databases that could well monitor patient results. In the Iraqi context, only a few studies have demonstrated the use of different trauma scores to predict outcomes in patients with trauma.

There is a significant research gap regarding the use of trauma scoring systems, especially TRISS, in Iraq. Most studies focus on descriptive outcomes rather than evaluating global trauma scores in the unique Iraqi context. Resource limitations, inconsistent pre-hospital care, and conflict-related injuries complicate the application of these systems. The lack of standardized trauma registries and data collection further limits the ability to improve trauma care and emergency services in Iraq.

ELIGIBILITY:
Inclusion Criteria:

* Trauma patients admitted to the emergency department of Al-Kadhimiya Teaching Hospital.
* Patients with adequate documentation of physiological and anatomical data are required for TRISS calculation.
* Trauma scoring (TRISS) completed within the first 6 hours of hospital arrival to ensure timely assessment.

Exclusion Criteria:

* Patients under 18 years, pregnant women, or those with conditions that alter standard trauma scoring or management.
* Non-trauma cases (e.g., medical emergencies, terminal illnesses) to ensure focus on trauma-specific outcomes.
* Patients with incomplete or missing data required for TRISS calculation.
* Patients declared dead on arrival or those not treated in the trauma and emergency department.
* Individuals refusing participation or withdrawing consent at any stage of the study.
* Patients transferred to or from another facility or enrolled in other studies that might affect scoring accuracy or outcomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of trauma patients presenting to the Emergency Department of Al-Kadhmia Teaching Hospital during the study period. These patients represent a diverse demographic and clinical profile, encompassing individuals with varying injury mechanisms, severities, and outcomes.
  The study specifically targets patients for whom trauma scoring systems, including the Trauma and Injury Severity Score (TRISS), can be applied reliably. This includes both blunt and penetrating trauma cases.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
In hospital mortality | In-Hospital Phase (average of 7-10 days through discharge); Post-Discharge Follow-Up: Day 7, Day 30
  Mortality (death) during hospitalization.
Accuracy Assessment of the Trauma and Injury Severity Score (TRISS) | the first 6 hours after ER admission
  A TRISS value close to 1 indicates a high probability of survival, while a value near 0 reflects a poor prognosis.

SECONDARY OUTCOMES:
Length of Hospitalization | Up to discharge, an average of 7-10 days
  The total duration of a patient's stay in the hospital, measured from the date of admission to the date of discharge. This includes all days spent in general wards, intensive care units (ICU), and other hospital departments as part of their treatment course.
Number of Participants Requiring ICU Admission | Up to discharge, an average of 7-10 days
  The requirement for admission to the intensive care unit (ICU) is determined by the presence of severe clinical deterioration, significant complications, or the need for advanced monitoring and life-support measures.
Need for Surgical Intervention | Up to discharge, an average of 7-10 days
  need for surgical intervention during a trauma patient's hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A. Hamdawi, Professor, Study Director — College Of Medicine - Nahrain University
Locations (1):
- College of Medicine - Al-Nahrain University, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haagsma JA, Graetz N, Bolliger I, Naghavi M, Higashi H, Mullany EC, Abera SF, Abraham JP, Adofo K, Alsharif U, Ameh EA, Ammar W, Antonio CA, Barrero LH, Bekele T, Bose D, Brazinova A, Catala-Lopez F, Dandona L, Dandona R, Dargan PI, De Leo D, Degenhardt L, Derrett S, Dharmaratne SD, Driscoll TR, Duan L, Petrovich Ermakov S, Farzadfar F, Feigin VL, Franklin RC, Gabbe B, Gosselin RA, Hafezi-Nejad N, Hamadeh RR, Hijar M, Hu G, Jayaraman SP, Jiang G, Khader YS, Khan EA, Krishnaswami S, Kulkarni C, Lecky FE, Leung R, Lunevicius R, Lyons RA, Majdan M, Mason-Jones AJ, Matzopoulos R, Meaney PA, Mekonnen W, Miller TR, Mock CN, Norman RE, Orozco R, Polinder S, Pourmalek F, Rahimi-Movaghar V, Refaat A, Rojas-Rueda D, Roy N, Schwebel DC, Shaheen A, Shahraz S, Skirbekk V, Soreide K, Soshnikov S, Stein DJ, Sykes BL, Tabb KM, Temesgen AM, Tenkorang EY, Theadom AM, Tran BX, Vasankari TJ, Vavilala MS, Vlassov VV, Woldeyohannes SM, Yip P, Yonemoto N, Younis MZ, Yu C, Murray CJ, Vos T. The global burden of injury: incidence, mortality, disability-adjusted life years and time trends from the Global Burden of Disease study 2013. Inj Prev. 2016 Feb;22(1):3-18. doi: 10.1136/injuryprev-2015-041616. Epub 2015 Dec 3. PMID 26635210
- [Result] Kelly JF, Ritenour AE, McLaughlin DF, Bagg KA, Apodaca AN, Mallak CT, Pearse L, Lawnick MM, Champion HR, Wade CE, Holcomb JB. Injury severity and causes of death from Operation Iraqi Freedom and Operation Enduring Freedom: 2003-2004 versus 2006. J Trauma. 2008 Feb;64(2 Suppl):S21-6; discussion S26-7. doi: 10.1097/TA.0b013e318160b9fb. PMID 18376168
- [Result] Penn-Barwell JG, Roberts SA, Midwinter MJ, Bishop JR. Improved survival in UK combat casualties from Iraq and Afghanistan: 2003-2012. J Trauma Acute Care Surg. 2015 May;78(5):1014-20. doi: 10.1097/TA.0000000000000580. PMID 25909424
- [Result] Lafta RK, Al-Nuaimi MA. National perspective on in-hospital emergency units in Iraq. Qatar Med J. 2013 Nov 1;2013(1):19-27. doi: 10.5339/qmj.2013.4. eCollection 2013. PMID 25003053
- [Result] Hussain AM, Lafta RK. Accidents in Iraq during the period of conflict (2003-2016). Qatar Med J. 2019 Dec 24;2019(3):14. doi: 10.5339/qmj.2019.14. eCollection 2019. PMID 31903321
- [Result] Champion HR, Copes WS, Sacco WJ, Lawnick MM, Keast SL, Bain LW Jr, Flanagan ME, Frey CF. The Major Trauma Outcome Study: establishing national norms for trauma care. J Trauma. 1990 Nov;30(11):1356-65. PMID 2231804
- [Result] Javali RH, Krishnamoorthy, Patil A, Srinivasarangan M, Suraj, Sriharsha. Comparison of Injury Severity Score, New Injury Severity Score, Revised Trauma Score and Trauma and Injury Severity Score for Mortality Prediction in Elderly Trauma Patients. Indian J Crit Care Med. 2019 Feb;23(2):73-77. doi: 10.5005/jp-journals-10071-23120. PMID 31086450
- [Result] Esme H, Solak O, Yurumez Y, Yavuz Y, Terzi Y, Sezer M, Kucuker H. The prognostic importance of trauma scoring systems for blunt thoracic trauma. Thorac Cardiovasc Surg. 2007 Apr;55(3):190-5. doi: 10.1055/s-2006-955883. PMID 17410508
- [Result] Wisner DH. History and current status of trauma scoring systems. Arch Surg. 1992 Jan;127(1):111-7. doi: 10.1001/archsurg.1992.01420010133022. No abstract available. PMID 1734842
- [Result] Imhoff BF, Thompson NJ, Hastings MA, Nazir N, Moncure M, Cannon CM. Rapid Emergency Medicine Score (REMS) in the trauma population: a retrospective study. BMJ Open. 2014 May 2;4(5):e004738. doi: 10.1136/bmjopen-2013-004738. PMID 24793256
- [Result] Karajizadeh M, Nasiri M, Yadollahi M, Zolfaghari AH, Pakdam A. Mortality Prediction from Hospital-Acquired Infections in Trauma Patients Using an Unbalanced Dataset. Healthc Inform Res. 2020 Oct;26(4):284-294. doi: 10.4258/hir.2020.26.4.284. Epub 2020 Oct 31. PMID 33190462
- [Result] Konesky KL, Guo WA. Revisiting traumatic cardiac arrest: should CPR be initiated? Eur J Trauma Emerg Surg. 2018 Dec;44(6):903-908. doi: 10.1007/s00068-017-0875-6. Epub 2017 Nov 25. PMID 29177620
- [Result] Mulvey HE, Haslam RD, Laytin AD, Diamond CA, Sims CA. Unplanned ICU Admission Is Associated With Worse Clinical Outcomes in Geriatric Trauma Patients. J Surg Res. 2020 Jan;245:13-21. doi: 10.1016/j.jss.2019.06.059. Epub 2019 Aug 5. PMID 31394403
- [Result] Todd KH, Lee T, Hoffman JR. The effect of ethnicity on physician estimates of pain severity in patients with isolated extremity trauma. JAMA. 1994 Mar 23-30;271(12):925-8. PMID 8120961
- [Result] Mondello S, Cantrell A, Italiano D, Fodale V, Mondello P, Ang D. Complications of trauma patients admitted to the ICU in level I academic trauma centers in the United States. Biomed Res Int. 2014;2014:473419. doi: 10.1155/2014/473419. Epub 2014 Jun 3. PMID 24995300
- [Result] Ramos-Pascua LR. Complications and trauma sequelae. Injury. 2018 Sep;49 Suppl 2:S1-S2. doi: 10.1016/j.injury.2018.06.045. Epub 2018 Jul 7. No abstract available. PMID 30097308
- [Result] Department of Error. Lancet. 2024 May 18;403(10440):1988. doi: 10.1016/S0140-6736(24)00824-9. Epub 2024 Apr 20. No abstract available. PMID 38648809
- [Result] Correction: Global injury morbidity and mortality from 1990 to 2017: results from the Global Burden of Disease Study 2017. Inj Prev. 2020 Oct;26(Supp 1):i165. doi: 10.1136/injuryprev-2019-043494corr1. Epub 2020 Sep 28. No abstract available. PMID 32989006
- See also: Injuries and violence. 19 June 2024 — https://www.who.int/news-room/fact-sheets/detail/injuries-and-violence